CLINICAL TRIAL: NCT04873570
Title: A Single Center, Open Label, Randomized, Single-dose, Two-period, Two-way Cross-over Study to Compare the Rate and Extent of Absorption of Mofest® 400mg (Moxifloxacin) Tablet With Avelox® 400mg (Moxifloxacin) Tablet in Healthy Pakistani Subjects.
Brief Title: Bioequivalence Study of Mofest® 400mg (Moxifloxacin) Tablet With Avelox® 400mg (Moxifloxacin) Tablet in Healthy Pakistani Subjects
Acronym: BE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Karachi (Other)
Collaborators: SAMI Pharmaceuticals (Pvt.) Ltd. (Industry); Center for Bioequivalence Studies and Clinical Research (Other)
Responsible Party: Principal Investigator, Dr. Muhammad Raza Shah, Professor, University of Karachi
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CB-034-MOX(M)-2020
Record Dates: First submitted 2021-04-28; First posted 2021-05-05 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Healthy Individuals; Bioequivalence Study
Keywords: Fluoroquinolone; Moxifloxacin; Bioequivalence; Pakistani Population
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Intervention Model Description: A single center, open label, randomized, single-dose, two-period, two-way cross-over study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test Group (Experimental): Subjects will be given one Mofest® 400mg (Moxifloxacin HCl) Tablet (1x400mg) manufactured by SAMI Pharmaceuticals (Pvt.) after at least 10 hours fast together with 240 mL of ambient temperature water at their scheduled dosing time-point. Blood samples will be taken up to 72.0 hours post-dose.
  Interventions: Drug: Moxifloxacin 400mg
- Reference Group (Active Comparator): Subjects will be given one Avelox® 400mg (Moxifloxacin HCl) Tablet (1x400mg), manufactured by Bayer HealthCare, after at least 10 hours fast together with 240 mL of ambient temperature water at their scheduled dosing time-point. Blood samples will be taken up to 72.0 hours post-dose.
  Interventions: Drug: Moxifloxacin 400mg

INTERVENTIONS:
Drug: Moxifloxacin 400mg — Moxifloxacin 400mg IR tablet

SUMMARY:
Single oral dose, of test and reference Tablet will be administered to healthy volunteers, after at least 10 hours fast together with 240 mL of ambient temperature water at their scheduled dosing time-points. Blood samples will be taken up to 72.0 hours post-dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged 18 to 55 years inclusive.
* Subjects with a body mass index (BMI) from 18.5 to 30 kg/m2.
* Subject is able to fast for 14 hours and consume standard meals.
* Subjects who are healthy as determined by routine physical examination, including vital sign monitoring (i.e., blood pressure, heart rate, and temperature), 12-Lead ECG, and safety laboratory analysis (i.e., hematology, blood biochemistry, and urinalysis) or viral serology as determined by the investigator.
* Subjects should have negative urine test for drugs of abuse (morphine & cannabinoids will be tested) and alcohol breath analysis at screening and prior to each check-in.
* Subjects who are able to, understand and sign the Informed Consent Form for Medical Screening during their screening visit and Participation Informed Consent Form on study check-In day.
* Subject agreed not to consume food or beverages including dairy products, tea, coffee, cola drinks, chocolates containing xanthine derivatives (including caffeine, theobromines, etc.) and/or poppy seeds (Khash khash) within 48 hours prior to drug administration until last blood draw in each study period.
* Subject agreed not to intake prescription drugs (especially amiodarone, carbamazepine, Antacids (aluminum and magnesium hydroxides) NSAIDS, digoxin and Blood thinners such as warfarin, etc.) within 14 days or 5 half-lives (whichever is longer) prior to first dose of study medicine.
* Subject agreed not to intake non-prescription drugs (OTC) within 14 days prior to first dose of study medicine.
* Subject agreed to discontinue vitamins, dietary and herbal supplements within 14 days prior to the first dose of study medication.
* Subject agreed not to consume grapefruit and/or its products within 14 days prior to the start of study.

Exclusion Criteria:

* Subjects who refused to sign Informed Consent Form.
* Subject not able to take medicine orally.
* Pregnant and lactating females.
* History of smoking ≥3 cigarette/day, alcoholism, and positive test for drug of abuse, heavy pan or gutka user as judged by teeth / mouth inspection.
* Subject has clinically relevant evidence of cardiovascular, gastrointestinal/hepatic, renal, psychiatric, respiratory, urogenital, hematological/immunologic, HEENT (head, ears, eyes, nose, throat), dermatological/connective tissue, musculoskeletal, metabolic/nutritional, drug hypersensitivity, allergy, endocrine, major surgery or other relevant diseases as revealed by medical history, physical examination, and laboratory assessments which may interfere with the absorption, distribution, metabolism or elimination of drugs or constitute a risk factor when taking study medication.
* Subjects known to be allergic to Moxifloxacin and/or other Quinolones antibiotics
* Subject who has received any other investigational drug within four weeks.
* Subject who has participated in any other clinical trials within 3 months.
* Donation or loss of more than 450 mL of blood within 3 months prior to the screening.
* History of any significant illness in the last four weeks which might confound in the result of the study or post additional risk in administrating Moxifloxacin to the subject.
* Subjects tested positive for syphilis (VDRL) or is known to have serum hepatitis or carrier of the Hepatitis B surface antigen (HBs Ag) or are carriers of antibodies to hepatitis C virus (anti-HCV) or to the human immunodeficiency virus (HIV-1 or HIV-2).

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pakistani Population
Enrollment: 38 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
maximum plasma concentration | up to 72 hours post dose
  maximum drug concentration in plasma after dose
Time to reach maximum plasma concentration | 0 to 72 hours post dose
  Time required for the drug to reach maximum plasma concentration
AUC | 0-72 hours
  Area under the time versus plasma drug concentration curve

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Muhammad R Shah, PhD, Principal Investigator — CBSCR, ICCBS, University of Karachi, Pakistan; Dr. Naghma Hashmi (Co-PI), PhD, Principal Investigator — CBSCR, ICCBS, University of Karachi, Pakistan
Locations (1):
- Center for Bioequivalence Studies and clinical research, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will only be available to other researchers upon reasonable request to PI keeping the participants' confidentiality intact.